CLINICAL TRIAL: NCT04968223
Title: Neural Correlates of Social Touch and Interoceptive Perception As Potential Biomarker for Impaired Social Functioning
Acronym: SPIRIT
Status: Completed | Type: Observational
Sponsor: University of Oldenburg (Other)
Collaborators: Danilo Postin, M.Sc. (Unknown)
Responsible Party: Principal Investigator, Dirk Scheele, Deputy Lab Head, University of Oldenburg
Other Study IDs: SPIRIT
Record Dates: First submitted 2021-06-11; First posted 2021-07-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: Biomarker-based prediction; Precision Psychiatry; Schizophrenia; Social functioning; Social Touch; Interoception; fMRI
MeSH Terms: conditions — Schizophrenia; Social Adjustment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples without DNA analysis, Urine samples without DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient Group: Patients with Schizophrenia
- Control Group: Healthy subjects without family history of psychotic illness

SUMMARY:
Recent studies have shown that certain biomarkers of schizophrenia could help to better assess the individual course of the disease and thus, contribute to more personalized treatment options. The aim of the SPIRIT study is to identify potential biomarkers for the prediction of disease-associated outcomes by investigating the neurobiological mechanisms of underlying schizophrenia-related dysfunctions.

DETAILED DESCRIPTION:
Alterations in psychosocial functioning are evident from the prodromal phase of schizophrenia and play a crucial role in its chronic course. While recent studies have demonstrated the predictive validity of structural changes in the brain anatomy of patients with schizophrenia, there is a lack of studies assessing the predictive value of disease-associated alterations in the functional brain activity for symptom severity and psychosocial functioning in schizophrenia.

In this longitudinal, observational study, 60 patients with schizophrenia and 40 healthy subjects without family history of psychotic illness will be recruited to investigate differences in behavioural, physiological, and neural correlates of social touch and interoceptive perception between participant groups. Participants' symptom severity and psychosocial functioning level will be examined by a wide range of behavioural, physiological, and neural methods. Potential biomarkers will be identified by estimating the predictive value of initially performed methods on follow-up re-examination of clinical and psychosocial outcomes. Neural readouts include structural and functional magnetic resonance imaging (fMRI) measurements. The fMRI tasks will probe the processing of social touch and interoceptive perception; additionally resting-state connectivity will be assessed. To further investigate pathological distortions of social touch and interoceptive perception, bodily touch allowance maps will be measured and participants will perform a heart-beat discrimination task. Psychometric questionnaires and semi-structured interviews will be used to capture symptom load and level of psychosocial functioning. Long-term effects will be assessed by online questionnaires and semi-structured interviews via phone call 3- and 6 months after initial assessments. The investigators hypothesize that differences in the neural response to social touch as well as in the neural patterns of interoceptive perception could serve as potential biomarkers for psychosocial deficits during the course of the illness. Furthermore, the inclusion of those biomarkers in predictive models could improve the prediction of disease progression and thus, contribute to personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to provide consent.
* Diagnosis of schizophrenia or schizoaffective disorder according to DSM-V
* Control group: No psychiatric or neurological illness.
* Fluent in German.

Exclusion Criteria:

* The participant does not fulfill requirements for MRI measurements according to safety guidelines.
* Acute suicidality.
* Current substance dependence.
* A history of head trauma or neurological illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In- and outpatients of the Department of Psychiatry, University of Oldenburg. Patients meeting the criteria for schizophrenia or schizoaffective disorder according to DSM-V will be included in the study. The patients' diagnosis will be verified via the structured clinical interview for DSM-V. Healthy subjects without family history of psychotic illness (control group). Control group will be matched to the patient sample.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Neural responses in a social touch task | One-time baseline assessment
  Participants will be measured with functional magnetic resonance imaging (fMRI) while they perceive different types of social and non-social touch
Behavioral responses in a social touch fMRI task | One-time baseline assessment
  Measured as behavioral ratings during the social touch fMRI task. During the social touch fMRI task, participants rate the comfort of the tactile stimuli on a visual analogue scale.
Neural responses in an interoception fMRI task | One-time baseline assessment
  Participants will be measured with functional magnetic resonance imaging (fMRI) while they perform an interoception task
Behavioral responses in an interoception fMRI task | One-time baseline assessment
  Measured by performance on the interoception task. During the interoception fMRI task, participants rate how intensely they perceived their heartbeat or their stomach on a visual analogue scale.
Changes in clinician-rated symptom severity between baseline and follow-ups | Baseline, 3 and 6 months follow- up after initial baseline assessment
  Measured by half-structured interviews (e.g. Positive and Negative Syndrome Scale (PANSS); range: 30-210; higher scores indicating more severe symptoms) for disease-related symptoms
Changes in self-reported symptom severity between baseline and follow-ups | Baseline, 3 and 6 months follow- up after initial baseline assessment
  Measured by self-evaluation questionnaires (e.g. Self-assessment of Negative Symptoms (SNS); range 1-20; higher scores indicating more severe symptoms) for disease-related symptoms
Changes in clinician-rated social-role functioning between baseline and follow-ups | Baseline, 3 and 6 months follow- up after initial baseline assessment
  Measured by the clinician-rated the social-role functioning scale (range: 1-10; higher scores indicating higher functioning)
Changes in self-reported social-role functioning levels between baseline and follow-ups | Baseline, 3 and 6 months follow-up after initial baseline assessment
  Measured by the self-evaluation questionnaires for social-role functioning (e.g. Social Network Index (SNI); range 1-12; higher scores indicating higher functioning)

SECONDARY OUTCOMES:
Bodily maps of social touch | One-time baseline assessment
  Measured as performance on a bodily maps computer task
Attitude towards social touch | One-time baseline assessment
  Measured by the self-evaluation questionnaire for social touch tolerance (e.g. Social Touch Questionnaire; range 0-4; higher scores indicating higher touch tolerance)
Interoceptive accuracy | One-time baseline assessment
  Measured as performance on a heartbeat discrimination task
Interoceptive awareness | One-time baseline assessment
  Measured by a self-evaluation questionnaire for interoceptive awareness (e.g. Multidimensional Assessment of Interoceptive Awareness (MAIA); range 0-5; higher scores indicating higher interoceptive awareness)
Blood parameter | One-time baseline assessment
  Measured by schizophrenia related, Nuclear Magnetic Resonance spectroscopy (NMR) based metabolomics
Urine parameter | One-time baseline assessment
  Measured by schizophrenia related, Nuclear Magnetic Resonance spectroscopy (NMR) based metabolomics
Neural activity at resting state | One-time baseline assessment
  fMRI will be performed to measure BOLD-signal while participants lay in the MRI-scanner with eyes open.
Structural connectivity measure | One-time baseline assessment
  fMRI will be performed to measure BOLD-signal while participants lay in the MRI-scanner with eyes open.

CONTACTS AND LOCATIONS:
Overall Officials: René Hurlemann, Prof., Principal Investigator — Department of Psychiatry, University of Oldenburg; Dirk Scheele, Dr., Principal Investigator — Department of Psychiatry, University of Oldenburg; Danilo Postin, M.Sc., Study Director — Department of Psychiatry, University of Oldenburg
Locations (1):
- Department of Psychiatry, University of Oldenburg, Bad Zwischenahn, Germany

IPD SHARING:
Plan to Share IPD: Undecided